CLINICAL TRIAL: NCT04240405
Title: Episodic Specificity Induction: Research of Its Explanatory Mechanisms and Application to Normal and Pathological Ageing.
Brief Title: Effects of Episodic Specificity Induction in Normal and Pathological Ageing.
Acronym: INSPE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19-0373
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Elderly people without cognitive impairment
- Amnestic type mild cognitive impairment patients (aMCI)
- Dysexecutive type mild cognitive impairment patients (dMCI)

SUMMARY:
Episodic Specificity Induction (ESI) is a short training that improves the production of episodic details during autobiographical recall in young and elderly people without cognitive impairment. But it remains to be determined 1) whether the mechanisms targeted by the ESI affect memory or executive functioning and 2) whether amnestic type (aMCI) or dysexecutive type (dMCI) mild cognitive impairment patients would benefit differently from this training, which has never been tested. By comparing the effect of the ESI on these patients, this would open up new perspectives for their symptomatic care.

ELIGIBILITY:
Inclusion Criteria:

The participant:

* has provided informed consent obtained in accordance with Good Clinical Practices.
* is affiliated to a social security system.
* speaks fluent French.
* is between 55 and 85 years of age.

For the participants of the control group:

* has a Montreal Cognitive Assessment (MoCA) score equal to or greater than 26;
* has neuropsychological assessment performance (RL/RI 16, D080, TMT, VOSP, Rey's figure) in the norm according to his socio-professional category and age, i.e. less than two deviating scores of -1 standard deviation or less than the 10th percentile per function.

For patients in the TCLa group:

* has at least two scores below the 10th percentile or below -1 standard deviation from the norm on neuropsychological assessment tests that assess memory, based on its socio-professional category and age;
* has less than two scores below the 10th percentile or less than -1 standard deviation from the norm in neuropsychological assessment tests that assess other functions. This is in accordance with the diagnostic criteria of Petersen (2004) and Jak and Bondi (2009).

For patients in the TCLd group:

* has focal executive dysfunction expressed by at least two scores less than the 10th percentile or less than -1 standard deviation from the norm in neuropsychological assessment tests that assess executive functions (TMT, Stroop, verbal fluences, free recall in memory), according to his socio-professional category and age;
* has less than two scores below the 10th percentile or less than -1 standard deviation from the norm on neuropsychological assessment tests that assess other functions (except for free memory reminders and language fluences). This is in accordance with the diagnostic criteria of Petersen (2004) and Jak and Bondi (2009).

Exclusion Criteria:

The participant:

* meets the criteria for a major neurocognitive disorder of the DSM-5.
* has a neurological disorder of infectious origin.
* has a psychiatric illness.
* has a severe uncompensated sensory deficit.
* is a substance abuser.
* has had chronic depression or anxiety that has not stabilized for 3 months.
* refuses to participate.
* is participating in another intervention research project.
* is placed under the protection of justice.
* refuses to sign the consent form.
* is unable to express its consent.
* consumed toxic substances or alcohol at the time of the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study looks at a population of adults between the ages of 55 and 85 and 3 types of sample of subjects extracted from this population :
  1. 24 elderly people without cognitive impairment
  2. 24 amnestic type mild cognitive impairment patients (aMCI)
  3. 24 dysexecutive type mild cognitive impairment patients (dMCI)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Average number of internal details | Day 0 (at inclusion)
  The participant sees 5 images evoking various events (e.g., a birthday, a restaurant) and describes for each one a related memory for 3 minutes. Each verbal production is recorded with a dictaphone, transcribed and then segmented into internal (episodic) or external (non-episodic) details according the coding procedure of Levine et al. (2002). The average number of internal details by autobiographical recall task is then calculated from these data.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Laboratoire d'Étude des Mécanismes Cognitifs, Bron
  - Centre Mémoire Ressources Recherche de Lyon, Institut du Vieillissement, Hôpital des Charpennes, Villeurbanne